CLINICAL TRIAL: NCT04668482
Title: Sweat Gland Function in Patients With Failed Back Surgery Syndrome, Treated With Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SWEAT2
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCS off (Experimental): SCS is switched off
  Interventions: Device: SCS is switched off
- SCS on (Experimental): SCS is switched on
  Interventions: Device: SCS is switched on

INTERVENTIONS:
Device: SCS is switched off — Spinal cord stimulator is switched off for 12 hours
  Arms: SCS off
Device: SCS is switched on — Spinal cord stimulator is functioning
  Arms: SCS on

SUMMARY:
This study is investigating sweat gland function during on and off states of the spinal cord stimulator, in patients with failed back surgery syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Diagnosis of FBSS (Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy) and currently being treated with spinal cord stimulation.
* Cognitive and language functioning enabling coherent communication between the examiner and the participant.

Exclusion Criteria:

* Patients with major psychiatric problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Sweat gland function by measuring Electrochemical Skin Conductances (ESC) | The change between the measurement while SCS is switched off and while SCS is switched on. Total study duration lasts one day.
  The investigators will examine the difference in sweat gland function between both measurements (SCS on versus SCS off), measured with the Sudoscan.

SECONDARY OUTCOMES:
Pain intensity scores using the Visual Analogue Scale | Two times on the same day; once while SCS is switched off and once while SCS is switched on. Total study duration lasts one day.
  Pain intensity score on that time on a Visual Analogue Scale (VAS) from zero (no pain) towards 10 cm (worst possible pain) for the pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium